CLINICAL TRIAL: NCT04337450
Title: A Randomised Non-inferiority Trial With Nested PK to Assess DTG/3TC Fixed Dose Formulations for the Maintenance of Virological Suppression in Children With HIV Infection Aged 2 to <15 Years Old
Brief Title: DTG/3TC Fixed Dose Formulations for the Maintenance of Virological Suppression in Children With HIV Infection Aged 2 to <15 Years Old
Acronym: D3 (Penta21)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: MRC CTU at UCL (Unknown); AMS-CMU/IRD (PHPT) (Unknown); Chris Hani Baragwanath Academic Hospital (Other); Durban International Clinical Research Site (Unknown); Hospital Universitario 12 de Octubre (Other); Prapokklao Hospital, Chantaburi (Unknown); Chiangrai Prachanukroh Hospital (Other); Nakornping Hospital (Other); Khon Kaen Hospital (Other Government); Kalasin Hospital (Other); Joint Clinical Research Center (Other); MU-JHU CARE (Other); Baylor College of Medicine (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Department of Clinical Pharmacy, University Medical Centre St Radboud, The Netherlands. (Other); Advanced Pathogens Diagnostics Unit, University College London Hospitals (Unknown); Centre for Health Economics, University of York (Unknown); Department of Molecular and Clinical Pharmacology, University of Liverpool (Unknown); St Mary's NHS Trust (Other Government); Chang Mai Univerity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3 (Penta21)
Record Dates: First submitted 2020-03-27; First posted 2020-04-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC (Active Comparator): Standard-of-care (SOC)
  Interventions: Drug: SOC
- DTG/3TC (Experimental): Dolutegravir (DTG) and lamivudine (3TC) (known as DTG/3TC)
  Interventions: Drug: Dolutegravir (DTG) and lamivudine (3TC)

INTERVENTIONS:
Drug: Dolutegravir (DTG) and lamivudine (3TC) — Children randomised to the DTG/3TC arm will receive once daily DTG/3TC fixed dose combination dispersible or film-coated tablets dosed using WHO weight bands criteria
  Arms: DTG/3TC
Drug: SOC — 2 nucleos(t)ide reverse transcriptase inhibitor (NRTI) and a third (anchor) drug (either an integrase strand transfer inhibitor (INSTI), a protease inhibitor (PI) or a non- nucleoside reverse transcriptase inhibitor (NNRTI)
  Arms: SOC

SUMMARY:
This study aims to find out whether treating children and young people living with HIV with two anti HIV medicines, dolutegravir and lamivudine, is safe and as effective as the three-medicine anti-HIV treatments currently used in routine practice.

DETAILED DESCRIPTION:
This study will include 370 children and young people aged 2 to less than 15 years old who are living with HIV and are being treated with anti-HIV medicines for the first time. Participants will be split into two groups, by chance, by a process called "randomisation". One group will continue to receive the anti-HIV medicines already taken according to country-specific routine practice. The second group will change to the new combination of medicine, dolutegravir and lamivudine (with the combination written usually as "DTG/3TC"). Depending on the weight, participants in the second group will be able take the new medicine either as one tablet a day or as a small number of dispersible tablets that are also taken once a day. All children and young people in the study will have regular clinic assessments that are at a similar frequency to the clinic visits that participants would have outside of the study. Blood tests will be performed to check that the medicine is safe and, at some visits, participants and their carers will also be asked to answer some questions on how they feel about taking their medicine. All children and young people will be followed until the last participant who joins the study has been in the study for 96 weeks.

After 96 weeks, children who were randomised to the DTG/3TC arm will enter the extended follow-up continuing to receive DTG/3TC.

ELIGIBILITY:
Inclusion Criteria for the Main trial:

1. HIV-1 infected children who are virologically suppressed for at least the last 6 months prior to enrolment
2. Aged 2 to <15 years old
3. Weight 6 kg or higher
4. Children on the same triple-drug PI/r, NNRTI or INSTI containing ART regimen for at least 3 months
5. Girls who have reached menarche must have a negative pregnancy test at screening and randomisation
6. Girls who are sexually active must be willing to adhere to highly effective methods of contraception
7. A parent or legal guardian is willing and able to give informed consent on behalf of the child as per national legislation and willing to adhere to the protocol
8. Participant is willing to give informed assent if the trial site clinician deems them old enough and able to understand the age-appropriate information about participation in the study

Inclusion Criteria for the Extended Follow up:

1. Participants remain on DTG/3TC at the end of the randomised phase, and in the opinion of the treating physician, derive ongoing benefit from DTG/3TC
2. Participants have no access to weight-appropriate DTG/3TC formulation via their national programme

Exclusion Criteria for the Main trial :

1. Any previous switch in ART regimen for virological, immunological or clinical treatment failure
2. Any changes in ART in the last 6 months for reasons other than due to child's growth, drug stock-outs, changes in country guidelines and treatment simplification
3. Evidence of previous resistance to 3TC or INSTI
4. Any prior use of regimens consisting of single or dual NRTIs with the exception of a course of zidovudine for PMTCT
5. Known allergy or contraindications to dolutegravir or lamivudine
6. Diagnosis of tuberculosis and on anti-tuberculosis treatment; children can be enrolled after successful tuberculosis treatment
7. Treatment of co-morbidities with drugs which have significant interactions with antiretroviral treatment, requiring dose adjustment of the study drugs (children can be enrolled after the illness resolves)
8. Randomisation visit more than 12 weeks after the most recent screening visit
9. Evidence of hepatitis B infection with no protective immunity against hepatitis B: participants positive for HBsAg or HBcAb and negative for HBsAb
10. Anticipated need for hepatitis C virus therapy with interferon-based regimen prior to the primary endpoint.
11. Screening ALT equal to 3 or more times the upper limit of normal AND bilirubin equal to 2 or more times the upper limit of normal (ALT ≥3xULN AND bilirubin ≥2xULN)
12. Screening ALT equal to 5 or more times the upper limit of normal ALT (≥5xULN)
13. Patients with severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
14. Screening creatinine clearance <50 mL/min/1.73m2
15. Patients aged ≥6 years at moderate or high risk of suicide as determined by Columbia-Suicide Severity Rating Scale (C-SSRS)
16. Girls who are pregnant or breastfeeding
17. Children who are in the legal custody of the State and do not have a parent or guardian able to provide informed consent on their behalf.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 386 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with confirmed viral rebound (defined as the first of two consecutive HIV-1 RNA ≥50c/mL) by week 96 | by Week 96

SECONDARY OUTCOMES:
Proportion of children with confirmed viral rebound (defined as the first of two consecutive HIV-1 RNA ≥50c/mL) by week 48 | by Week 48
Proportion of children with confirmed HIV-1 RNA ≥50c/mL at weeks 48 and 96 (modified FDA snapshot) | at Week 48 and 96
Proportion of children with HIV-1 RNA ≥50c/mL at weeks 24, 48 and 96 (including blips and confirmed measures ≥50c/mL) | at Week 24, 48 and 96
New resistance-associated mutations in those with confirmed HIV-1 RNA ≥50c/mL | by Week 96
Time to any new or recurrent WHO 3 or WHO 4 event or death | through study completion, up to 5 years
Change in CD4 (absolute and percentage) from baseline to weeks 24, 48 and 96 | Week 24, 48 and 96
Incidence of serious adverse events, grade 3 and 4 clinical and laboratory adverse events | through study completion, up to 5 years
Incidence of adverse events leading to discontinuation or modification of the treatment regimen | through study completion, up to 5 years
Proportion of children with a change in ART for toxicity or switch to second-line | through study completion, up to 5 years
Change in blood lipids from baseline to weeks 48 and 96 | Week 48 and 96
Change in creatinine clearance estimated using bedside-Schwartz to weeks 48 and 96 | Week 48 and 96

CONTACTS AND LOCATIONS:
Locations (14):
- South Africa (3):
  - King Edward VIII Hospital, Durban
  - PHRU Klerksdorp, Klerksdorp
  - PHRU, Soweto
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Thailand (4):
  - Prapokklao Hospital, Chanthaburi
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Khon Kaen Hospital, Khon Kaen
- Uganda (3):
  - Baylor, Kampala
  - Joint Clinical Research Centre, Kampala
  - MUJHU, Kampala
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Great Ormand Street Hospital, London
  - St. Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turkova A, Chan MK, Kityo C, Kekitiinwa AR, Musoke P, Violari A, Variava E, Archary M, Cressey TR, Chalermpantmetagul S, Sawasdichai K, Ounchanum P, Kanjanavanit S, Srirojana S, Srirompotong U, Welch S, Bamford A, Epalza C, Fortuny C, Colbers A, Nastouli E, Walker S, Carr D, Conway M, Spyer MJ, Parkar N, White I, Nardone A, Thomason MJ, Ferrand RA, Giaquinto C, Ford D; D3 trial team. D3/Penta 21 clinical trial design: A randomised non-inferiority trial with nested drug licensing substudy to assess dolutegravir and lamivudine fixed dose formulations for the maintenance of virological suppression in children with HIV-1 infection, aged 2 to 15 years. Contemp Clin Trials. 2024 Jul;142:107540. doi: 10.1016/j.cct.2024.107540. Epub 2024 Apr 16. PMID 38636725
- [Derived] Botha JC, Byott M, Spyer MJ, Grant PR, Gartner K, Chen WX, Burton J, Bamford A, Waters LJ, Giaquinto C, Turkova A, Vavro CL, Nastouli E. Sensitive HIV-1 DNA Pol Next-Generation Sequencing for the Characterisation of Archived Antiretroviral Drug Resistance. Viruses. 2023 Aug 25;15(9):1811. doi: 10.3390/v15091811. PMID 37766218
- See also: Related Info — https://penta-id.org/
- See also: Related Info — https://www.ctu.mrc.ac.uk/